CLINICAL TRIAL: NCT04435223
Title: Lipid Metabolism in COVID-19 Severe Pneumonia Compared With Severe Pneumonia Caused by Other Pathogen
Acronym: COVIDOLIP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NGUYEN AOIc 2020
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Severe Pneumonia; Severe Pneumonia Due to Other Pathogene
MeSH Terms: interventions — Biological Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 severe pneumonia
  Interventions: Biological: biological assays in particular on the lipid metabolism
- Severe pneumonia due to other pathogene
  Interventions: Biological: biological assays in particular on the lipid metabolism

INTERVENTIONS:
Biological: biological assays in particular on the lipid metabolism — bioassays carried out on samples already collected and conserved

SUMMARY:
SARS-COV 2 infection might be responsible for sever pneumonia. Obesity seems to be a risk factor for severe SARS-COV 2 pneumonia. Lipid metabolism alteration are described with both obesity and sepsis. The aim of the present study was to describe association between lipid metabolism, obesity, sepsis inflammation and clinical outcome in COVID-19 patient with severe pneumonia compared with severe pneumonia caused by other pathogenes.

ELIGIBILITY:
Inclusion Criteria:

* 2 of the following criteria: Cough/ Dyspnea/ Spitting/ Thoracic pain/ Hyperthermia (>=38 °C) Hypothermia (< 35°C) AND new radiologic pulmonary infiltrate
* At admission or within 48 hours following hospital admission
* With 2 qSOFA criteria: MAP =< 100 mmHg, Respiratory Rate >= 22, Glasgow score < 15 OR on mechanical ventilation OR under vasopressor
* Age > 18
* affiliated to social security

Exclusion Criteria:

* Pregnancy
* immunodepression
* Pathology known to cause severe lymphopenia
* hospitalisation within 3 month before inclusion AND sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with pneumopathy
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Cholesterol concentration | Within 48 hours following hospital admission

SECONDARY OUTCOMES:
LDL cholesterol / HDL cholesterol/ Lipoprotein size and composition/ Non esterified Fatty acid/ Triglyceridemia/ CETP and PLTP activity/ apolipoprotein canceration/ lipid peroxidation/ Pro and anti inflammatory profile. | Within 48 hours following hospital admission
  Ventilator free days (28 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Nguyen M, Bourredjem A, Piroth L, Bouhemad B, Jalil A, Pallot G, Le Guern N, Thomas C, Pilot T, Bergas V, Choubley H, Quenot JP, Charles PE, Lagrost L, Deckert V, de Barros JP, Guinot PG, Masson D, Binquet C, Gautier T, Blot M; Lymphonie study group. High plasma concentration of non-esterified polyunsaturated fatty acids is a specific feature of severe COVID-19 pneumonia. Sci Rep. 2021 May 24;11(1):10824. doi: 10.1038/s41598-021-90362-9. PMID 34031519